CLINICAL TRIAL: NCT02184559
Title: Postoperative Analgesia After Caesarean Section Under ALR: TAP Block Versus Catheter Scar Infiltration
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-005690-23; 2011-38 (Other: AP HM)
Record Dates: First submitted 2014-06-25; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Scheduled Caesarian Section
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP block (Experimental)
  Interventions: Drug: Ropivacaine
- infiltration continues (Active Comparator)
  Interventions: Device: The infiltration continues catheter

INTERVENTIONS:
Drug: Ropivacaine — comparaison of two methods of administration for analgesia using the same drugs in the same indication after Caesarean section
  Arms: TAP block
Device: The infiltration continues catheter
  Arms: infiltration continues

SUMMARY:
The purpose of the multimodal postoperative analgesia is to improve the quality of analgesia and reduce side effects of morphine (nausea, vomiting, sedation, urinary retention, respiratory depression ...). In the case of caesarean sections, the quality of analgesia allows one hand to improve the mother-child relationship and the quality of breastfeeding, the other to reduce the risk of postpartum depression and chronic pain . Two methods of administration of local anesthetics have been proven effective for analgesia of the abdominal wall under umbilical: The Transversus Abdominal Block Plan (TAP Block) and infiltration of the scar continues operating. The TAP block was performed under ultrasound guidance by the anesthesiologist after the intervention in a single injection of local anesthetic in the abdominal wall and has a period of limited and variable. The infiltration continues catheter is placed by the surgeon before closing the wound and allows the infusion of local anesthetics for 48 hours.

The purpose of this study was to compare morphine consumption between both techniques, and the quality of analgesia and side effects of morphine

ELIGIBILITY:
Inclusion Criteria:

* Woman whose age is 18 years
* Encircled Woman requiring a scheduled(programmed) caesarian, under spinal anesthesia or died combined(organized) spinal anesthesia
* Woman ASA I and II
* Term = 37 LIMITED COMPANIES
* Woman primipare or not
* Woman having signed an informed consent writes and making a commitment to respect the instructions of the protocol

Exclusion Criteria:

* Minor Woman
* Woman presenting a contraindication to the anesthesia périmédullaire: constitutional or acquired disorders(confusions) of the haemostasis, the allergy in the local anesthetics, the infectious context (hypertherm > 38.5 ° C)
* Woman presenting an intolerance or an allergy known about the morphine in the paracetamol or in AIN
* The surgical histories of laparotomy
* The morbid obesity BMI > 35
* Dysgravidies
* Woman not being affiliated to the national insurance scheme
* Woman under legal protection
* Woman not having signed an informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-08 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Consumption morphinize | 48 hours
  the cosumption of morphinize is collected since the first hours of comsumption to the 48 th hours

SECONDARY OUTCOMES:
Analgesic efficiency | 48 hours
  the Score of pain measured by simple numerical rating scales start the first hours one asks for a complementary analgesia to the 48 th hours

CONTACTS AND LOCATIONS:
Overall Officials: loic MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France